CLINICAL TRIAL: NCT05854524
Title: Exploring the Biological Basis for Exercise Neuroprotection in Parkinson's Disease
Brief Title: Exercise Neuroprotection in Parkinson's Disease
Acronym: PDex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Merrill Landers, Professor and Chair, University of Nevada, Las Vegas
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: UNLVPT PDex2023.01
Record Dates: First submitted 2023-04-13; First posted 2023-05-11 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: Exercise; Inflammation; Physical activity; Neuroprotection
MeSH Terms: conditions — Parkinson Disease; Motor Activity; Inflammation | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a cross-over design with two arms (Parkinson Disease and healthy control) and two conditions (low and high intensity aerobic exercise). The interventions for this Phase II trial are two different intensities of aerobic exercise.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and the outcomes assessors will be blinded to the main purpose and aims of the study. Additionally, both conditions are aerobic exercise conditions of different intensities so they will clearly know that they are exercising but will not know the main purpose behind the two different intensities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parkinson Disease (Active Comparator): Participants diagnosed with Parkinson disease (PD) will the main arm of the study and will be compared to the control group.
  Interventions: Procedure: Aerobic exercise
- Control (Active Comparator): Older, adults who are age- and sex-matched to the PD participants.
  Interventions: Procedure: Aerobic exercise

INTERVENTIONS:
Procedure: Aerobic exercise — The intervention is exercise and there are no drugs or devices used in this trial. The exercise consists of two intensity levels of a 30-minute aerobic exercise intervention with both arms crossing over to both conditions: low intensity exercise (60-70% of estimated maximum heart rate (EMRH)) and moderate-vigorous intensity exercise (75-85% of EMHR).

SUMMARY:
The purpose of this study is to explore the relationships of exercise on inflammation in the body of older adults and people with Parkinson's disease (PD). This is important research for older adults but is especially important for people with PD because neuroinflammation is the main pathological mechanism that is responsible for neuron cell death in this neurodegenerative disease. As PD is a progressive disease, halting or slowing the degeneration is an important research target. Halting or slowing the disease progress is known as neuroprotection. Exercise is an attractive therapeutic treatment for people with PD as it has a lot of multi-systemic benefits, but also there is a lot of evidence to suggest that it helps improve symptoms and slow the progression of the disease. Exercise has been theorized to decrease inflammation and, therefore, has a lot of promise as a neuroprotective agent in slowing or halting the degeneration in PD. Unfortunately, there is not a lot of research that has looked into the effect of exercise on the biological processes of inflammation. Thus, the purpose of this study is to investigate the biological evidence that underlies the positive effect of exercise in people with PD.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disease, affecting an estimated 4 million individuals and 1% of those over the age of 60. The pathologic hallmark of PD are Lewy bodies in neurons and these inclusion bodies are largely made up of misfolded α-synuclein. These α-synuclein inclusion bodies cause mitochondrial respiratory dysfunction which results in reactive oxygen species causing oxidative stress; this, in turn, leads to more aggregation of α-synuclein and a vicious cycle ensues. Ultimately, this vicious cycle results in dopaminergic neuron cell death causing a decrease in dopamine in the nigrostriatal pathway. Mitochondrial dysfunction and subsequent oxidative stress are also caused by environmental toxins (e.g., trichloroethylene, paraquat) and neuroinflammation, both of which are theorized to play a prominent role in PD pathology. Because of this, neuroprotective strategies in PD have focused on limiting exposure to environmental toxins and, more importantly, decreasing pro-inflammatory mechanisms.

Evidence has been accumulating that exercise improves symptoms and quality of life and is neuroprotective in PD. In one meta-analysis, they found that regular exercise delays the progression of PD motor symptoms, mobility, and balance deterioration. Another meta-analysis reported a reduced risk for developing PD in the pre-clinical phase for those performing moderate to vigorous exercise. Another meta-analysis showed a 40% risk reduction in developing PD for people regularly performing moderate to vigorous activity aged 35-39 or within the previous ten years. Based on these findings, it can be reasonably deduced that moderate to vigorous exercise prior to PD diagnosis is neuroprotective. Moreover, exercise may also slow the progression of degeneration after PD diagnosis.

A prominent theory underlying neuroprotection in PD is that exercise may mitigate the pro-inflammatory milieu thereby protecting and slowing the progressive loss of dopaminergic neurons. Various chemical mediators, antioxidant agents, and cytokines have been shown to play a role in the development, progression, and severity of PD, including interleukin 6 (IL-6) and 10 (IL-10), tumor necrosis factor (TNF), and the interferon gamma family (IFNγ). Some of these chemicals are anti-inflammatory and some are pro-inflammatory. While these are some of the most commonly studied cytokines, there are many others that are understudied in PD and they may also contribute to the internal state of inflammation in PD. Therefore, it is important to examine the collective blend of these cytokines and chemokines to understand the inflammatory milieu in PD as a result of acute and chronic exercise. While regular exercise may be neuroprotective in PD by reducing oxidative stress, the release of antioxidant enzymes via exercise (superoxide dismutase (SOD), glutathione peroxidase, catalase) may also contribute to an overall decrease in the state of inflammation in PD.

Another group of compounds theorized to play a role in the mitigation of PD progression are the neurotrophins (e.g., brain-derived neurotrophic factor (BDNF), vascular endothelial growth factor (VEGF), glial cell line-derived neurotrophic factor (GDNF)). All three of the aforementioned neurotrophins are activity-dependent meaning they increase as a result of exercise. GDNF and BDNF have received the most attention and are theorized to aid in neuroregeneration and neuroprotection in PD by protecting dopaminergic neurons. There are decreased levels of BDNF in the dopaminergic nigrostriatal pathways in people with PD (PwP). A reduction in the bioavailability of dopamine compounded by a decrease in BDNF has been shown to be associated with PD signs (movement dysfunction, resting tremor, and bradykinesia). Additionally, BDNF may also be related to an anti-inflammatory milieu in PD thereby highlighting the need to investigate the cytokines and neurotrophins together. Lastly, VEGF may indirectly impact neuroprotection in PD by improving blood supply (angiogenesis) and synaptic activity.

Thus, there are three possible mechanisms that are theorized to underlie the disease modifying effects of exercise in PD: decreasing the inflammatory milieu via cytokines, decreasing the inflammatory milieu via antioxidant enzymes, and improved neuroprotection of neurons via neurotrophins. Currently, it is not understood if one of these methods predominates or if it is the combination of these mechanisms that underlie neuroprotection. Theoretically, all three mechanisms may slow the progression of PD by breaking up the vicious cycle of α-synuclein aggregation, mitochondrial toxicity, and oxidative stress. These purported mechanisms warrant further research attention. Importantly, there are no studies to our knowledge that have looked at all three mechanisms together in one study. Since there are interrelationships among the three mechanisms it makes sense to explore these in more detail. Importantly, it is not known how these mechanisms respond to different doses of exercise. Therefore, this study will examine the relationship of exercise dose to these mechanisms to gain greater insight into neuroprotection in PD. The following are the specific aims of this study:

Primary Aim 1 (exercise and inflammatory milieu): To determine if there is an association between current exercise/physical activity habits and levels of cytokines, antioxidant enzymes, and neurotrophins after controlling for PD progression, age, sex, body mass index, inflammatory-related genotypes, and number of comorbidities.

Hypothesis 1: PwP who are regular exercisers will have less inflammation (more anti-inflammatory cytokines and/or fewer pro-inflammatory cytokines) and higher levels of antioxidant enzymes and neurotrophins compared to those who are not regular exercisers.

Primary Aim 2 (inflammatory milieu comparison to controls): To determine if there is a difference between PwP and healthy controls on levels of cytokines, antioxidant enzymes, and neurotrophins after controlling for age, sex, body mass index, inflammatory-related genotypes, and number of comorbidities.

Hypothesis 2: PwP will have higher levels of more inflammation and lower levels of antioxidant enzymes and neurotrophins compared to healthy, age-matched controls.

Primary Aim 3 (exercise dose and biomarkers): To determine if there is a difference before and after 30 minutes of aerobic exercise at 60-70% and 75-85% of the estimated maximum heart rate (EMHR) in PwP and healthy, age-matched controls.

Hypothesis 3: There will be an interaction (e.g., different slope of pro- and anti-inflammatory cytokines) between prior level of exercise (regular exercisers versus non-regular exercisers using the Centers for Disease Control (CDC) 150 minutes of regular exercise per week), exercise intensity (60-70% and 75-85% of EMHR), and status (PwP and control) on the change in inflammation, antioxidant enzymes, and neurotrophins.

Primary Aim 4 (biomarkers in PD): To determine which of an array of biomarkers is most associated with PD compared to controls and which of those biomarkers is the most associated with exercise and PD progression (MDS-UPDRS score divided by years since diagnosis).

Hypothesis 4: Among an array of markers, the investigators expect to see the difference between PwP and controls for the following: cytokines, antioxidant enzymes, and neurotrophins.

Hypothesis 5: Among an array of markers, the investigators expect to see the greatest changes before and after higher intensity exercise in PwP in the following: cytokines, antioxidant enzymes, and neurotrophins.

ELIGIBILITY:
Inclusion criteria for PwP:

* 30-85 years old
* Neurologist-diagnosed PD
* Able to participate in 30 minutes of continuous moderate aerobic exercise with 2-3 short breaks per self-report.

Inclusion criteria for controls:

* 30-85 years old
* No major medical diagnoses
* Able to participate in 30 minutes of continuous moderate aerobic exercise with 2-3 short breaks per self-report.

Exclusion Criteria for both PD group and controls:

* Diagnoses, identified by self-report, that would preclude exercise participation (e.g., heart arrhythmias, uncontrolled blood pressure, exercise-induced asthma).
* Those not deemed ready for exercise participation. Participants will be screened for exercise participation using the Physical Activities Readiness Questionnaire + which is used as a screening tool for all ages to identify risk factors that would clear someone for participation in moderate physical exercise.
* Those with dementia will be excluded because there are self-report questionnaires in this study. This will be identified using the Montreal Cognitive Assessment and a score at or below a 21. Participants with mild cognitive impairment and no impairment will be included.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Exercise and inflammatory milieu | Baseline measurement only
  International Physical Activity Questionnaire (IPAQ) and blood serum levels of the following: interleukin-6 (IL-6), tumor necrosis factor alpha (TNF), interleukin-1β (IL-1β), interleukin-2 (IL-2), interleukin-10 (IL-10), c-reactive protein (CRP), RANTES, BDNF, VEGF, nerve growth factor (NGF), GDNF, Superoxide dismutase, catalase, glutathione peroxidase, total antioxidant capacity
Inflammatory milieu comparison to controls | Baseline measurement only
  Blood serum levels of the following: IL-6, TNF, IL-1β, IL-2, IL-10, CRP, RANTES, BDNF, VEGF, NGF, GDNF, Superoxide dismutase, catalase, glutathione peroxidase, total antioxidant capacity
Exercise dose and biomarkers | 30 minutes prior to the exercise (pre measurement) and 30 minutes after completing the 30-minute aerobic exercise condition (post measurement) . Both conditions are separated by one week.
  Change in blood serum levels of the following for the two different exercise conditions: IL-6, TNF, IL-1β, IL-2, IL-10, CRP, RANTES, BDNF, VEGF, NGF, GDNF, Superoxide dismutase, catalase, glutathione peroxidase, total antioxidant capacity, deglycase (DJ-1) protein, nonenzymatic antioxidants (Glutathione, Vitamin A, Vitamin C, Vitamin E).
Biomarkers in Parkinson Disease | 30 minutes prior to the exercise (pre measurement) and 30 minutes after completing the 30-minute aerobic exercise condition (post measurement) . Both conditions are separated by one week
  Change in blood serum levels of the following for people with Parkinson's disease and older adults: IL-6, TNF, IL-1β, IL-2, IL-10, CRP, RANTES, BDNF, VEGF, NGF, GDNF, Superoxide dismutase, catalase, glutathione peroxidase, total antioxidant capacity, DJ-1 protein, nonenzymatic antioxidants (Glutathione, Vitamin A, Vitamin C, Vitamin E).

CONTACTS AND LOCATIONS:
Overall Officials: Merrill Landers, DPT, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- Gait and Balance Laboratory, 217 Bigelow Health Sciences Building, UNLV, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
There is not plan to share data with other researchers at this time.

REFERENCES:
- [Background] Chao Y, Wong SC, Tan EK. Evidence of inflammatory system involvement in Parkinson's disease. Biomed Res Int. 2014;2014:308654. doi: 10.1155/2014/308654. Epub 2014 Jun 24. PMID 25050341
- [Background] Kim R, Kim HJ, Kim A, Jang M, Kim A, Kim Y, Yoo D, Im JH, Choi JH, Jeon B. Peripheral blood inflammatory markers in early Parkinson's disease. J Clin Neurosci. 2018 Dec;58:30-33. doi: 10.1016/j.jocn.2018.10.079. Epub 2018 Oct 24. PMID 30454693
- [Background] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886
- [Background] Zhang M, Li F, Wang D, Ba X, Liu Z. Exercise sustains motor function in Parkinson's disease: Evidence from 109 randomized controlled trials on over 4,600 patients. Front Aging Neurosci. 2023 Feb 14;15:1071803. doi: 10.3389/fnagi.2023.1071803. eCollection 2023. PMID 36865410
- [Background] Fang X, Han D, Cheng Q, Zhang P, Zhao C, Min J, Wang F. Association of Levels of Physical Activity With Risk of Parkinson Disease: A Systematic Review and Meta-analysis. JAMA Netw Open. 2018 Sep 7;1(5):e182421. doi: 10.1001/jamanetworkopen.2018.2421. PMID 30646166
- [Background] Xu Q, Park Y, Huang X, Hollenbeck A, Blair A, Schatzkin A, Chen H. Physical activities and future risk of Parkinson disease. Neurology. 2010 Jul 27;75(4):341-8. doi: 10.1212/WNL.0b013e3181ea1597. PMID 20660864
- [Background] Palasz E, Wysocka A, Gasiorowska A, Chalimoniuk M, Niewiadomski W, Niewiadomska G. BDNF as a Promising Therapeutic Agent in Parkinson's Disease. Int J Mol Sci. 2020 Feb 10;21(3):1170. doi: 10.3390/ijms21031170. PMID 32050617
- [Background] da Silva PG, Domingues DD, de Carvalho LA, Allodi S, Correa CL. Neurotrophic factors in Parkinson's disease are regulated by exercise: Evidence-based practice. J Neurol Sci. 2016 Apr 15;363:5-15. doi: 10.1016/j.jns.2016.02.017. Epub 2016 Feb 10. PMID 27000212
- [Background] Zoladz JA, Majerczak J, Zeligowska E, Mencel J, Jaskolski A, Jaskolska A, Marusiak J. Moderate-intensity interval training increases serum brain-derived neurotrophic factor level and decreases inflammation in Parkinson's disease patients. J Physiol Pharmacol. 2014 Jun;65(3):441-8. PMID 24930517